CLINICAL TRIAL: NCT00417209
Title: A Randomized, Open Label Multi-Center Study Of Single Agent Larotaxel (XRP9881) Compared To Continuous Administration of 5-FU For The Treatment Of Patients With Advanced Pancreatic Cancer Previously Treated With A Gemcitabine-Containing Regimen
Brief Title: Larotaxel Compared To Continuous Administration of 5-FU in Advanced Pancreatic Cancer Patients Previously Treated With A Gemcitabine-Containing Regimen
Acronym: PAPRIKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6596; EUDRACT: 2006-003086-14
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Neoplasms
Keywords: advanced pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — larotaxel; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Larotaxel (XRP9881) (Experimental)
  Interventions: Drug: Larotaxel (XRP9881)
- 5-Fluorouracil or capecitabine (Active Comparator): Each Investigator must choose either IV 5-FU or oral capecitabine regimen before the first participant begins the study and has to consistently use the chosen regimen throughout the study for all participants treated at her/his site.
  Interventions: Drug: 5-Fluorouracil; Drug: Capecitabine

INTERVENTIONS:
Drug: Larotaxel (XRP9881) — administered as a 1-hour IV infusion on Day 1 of every 3 weeks (q3w)
  Arms: Larotaxel (XRP9881)
Drug: 5-Fluorouracil — administered as IV infusion from Day 1 to Day 4
  Arms: 5-Fluorouracil or capecitabine
Drug: Capecitabine — administered orally from Day 1 to Day 14 q3w
  Arms: 5-Fluorouracil or capecitabine

SUMMARY:
The purpose of this study is to compare the efficacy and the safety Larotaxel administered as single agent every 3 weeks to continuous administration of 5-FU every 3 weeks, in patients with advanced pancreatic cancer (non operable in a curative intent, locally recurrent or metastatic) previously treated with gemcitabine based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (non operable in a curative intent, locally recurrent or metastatic disease) Cytologically or histologically proven epithelial cancer (adenocarcinoma) of the exocrine pancreas.
* Patient must be previously treated with a systemic gemcitabine based regimen
* Adequate bone marrow, kidney and liver functions

Exclusion Criteria:

* ECOG performance status (PS) of 2-3-4.
* Prior locoregional radiotherapy for pancreatic cancer.
* Symptomatic brain metastases or leptomeningeal disease.
* Any serious intercurrent infections, uncontrolled cardiac or gastro-intestinal diseases.
* Other concurrent malignancy
* Other protocol-defined exclusion/inclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) defined as the time interval from the date of randomization to the date of death due to any cause | study period

SECONDARY OUTCOMES:
Progression free survival (PFS); Overall Response Rate (proportion of patients with confirmed RECIST-defined complete response (CR) or partial response (PR); clinical benefit based on the measurement of tumor related symptoms; | study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (21):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Lima, Peru
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Brastislava, Slovakia
- Sanofi-Aventis Administrative Office, Madrid, Spain
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom